CLINICAL TRIAL: NCT02811562
Title: Learning Curves of Intubation for Simulated Difficult Airway Scenarios by Manikin: Comparison of Combined Pentax Airwayscope-fiberoptic Bronchoscope and Fiberoptic Bronchoscope Alone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, DAE HEE KIM, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AJIRB-DEV-EXP-16-116
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Difficult Airway

ARMS (2):
- fiberoptic bronchoscope (Active Comparator): Tracheal intubation in manikin using fiberoptic bronchoscope
  Interventions: Device: manikin; Device: fiberoptic bronchoscope
- fiberoptic bronchoscope with pentax-airwayscope (Experimental): Tracheal intubation in manikin using fiberoptic bronchoscope with pentax-airwayscope
  Interventions: Device: manikin; Device: fiberoptic bronchoscope; Device: pentax-airwayscope

INTERVENTIONS:
Device: manikin
Device: fiberoptic bronchoscope
Device: pentax-airwayscope
  Arms: fiberoptic bronchoscope with pentax-airwayscope

SUMMARY:
Acquisition of knowledge and skills pertinent to the use of fibreoptic endoscopy is an important part of training in various medical and surgical specialties such as anesthesiology, emergency medicine, otolaryngology, and pulmonary medicine. It has been shown that there is a wide variation in the learning curves of residents and the number of attempts to achieve proficiency in performing upper airway endoscopy. recently, combined use of fiberoptic bronchoscope and videolaryngoscope has been suggested to be a good alternative. So, the aim of this study is to compare the number of attempt to achieve proficiency using fiberoptic bronchoscope alone or fiberoptic bronchoscope with Pentax-AWS.

ELIGIBILITY:
Inclusion Criteria:

* resident in Department of anesthesiology

Exclusion Criteria:

* resident who has an experience of successful fiberoptic bronchoscopic intubation in difficult case

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
trial number to achieve 'proficient' in terms of cumulative sum analysis | up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hee Kim, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou universiry hospital, Suwon, Gyeonggi-do, South Korea